CLINICAL TRIAL: NCT01426919
Title: A Prospective Clinical Evaluation of Biomarkers of Traumatic Brain Injury
Brief Title: Evaluation of Biomarkers of Traumatic Brain Injury
Acronym: ALERT-TBI
Status: Completed | Type: Observational
Sponsor: Banyan Biomarkers, Inc (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ATO-06
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Head Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected traumatic brain injury with head CT
  Interventions: Other: Head CT scan and blood draw within 12 hours of injury

INTERVENTIONS:
Other: Head CT scan and blood draw within 12 hours of injury

SUMMARY:
The primary objective of this study is to evaluate the utility of the Banyan UCH-L1/GFAP Detection Assay as an aid in the evaluation of suspected traumatic brain injury (Glasgow Coma Scale score 9-15) in conjunction with other clinical information within 12 hours of injury to assist in determining the need for a CT scan of the head.

ELIGIBILITY:
Inclusion Criteria:

* subject is at least 18 years of age at screening
* suspected traumatically induced head injury as a result of insult to the head from external force
* GCS 9-15 at time of informed consent
* workup includes head CT scan as part of clinical emergency care within 3 hours of presenting and within 12 hours of injury
* blood sample collected within 3 hours of presenting and within 12 hours of injury
* subject or legal representative is willing to undergo informed consent

Exclusion Criteria:

* participating in an interventional, therapeutic clinical study that may affect the results of this study (an observational study acceptable)
* time of injury cannot be determined
* primary diagnosis of ischemic or hemorrhagic stroke
* venipuncture not feasible
* a condition precluding entry into the CT scanner
* subject has a neurodegenerative disease or other neurological disorder including dementia, Parkinson's disease, multiple sclerosis, seizure disorder, brain tumors, and history of neurosurgery, stroke or TIA within the last 30 days
* administration of blood transfusion after head injury and prior to study blood draw
* subject is otherwise determined by the Investigator to be unsuitable for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for study participation will be over the age of 18 and present to the health care facility with a head injury at a time such that sample collection can be completed within 12 hours of injury. Subjects who will be permitted into the study include those who will meet all the inclusion criteria and will have none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2011 (Actual)
Dates: Start 2012-12; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Correlation of assay result with absence of acute intracranial lesions | Day 1

CONTACTS AND LOCATIONS:
Locations (24):
- United States (17):
  - University of California San Diego, San Diego, California
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Wayne State University - Detroit Receiving Hospital, Detroit, Michigan
  - Wayne State University - Sinai Grace Hospital, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University Medical Center Brackenridge, Austin, Texas
  - Baylor College of Medicine/Ben Taub General Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Carilion New River Valley, Christiansburg, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
- Germany (5):
  - Charité Universitätsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Charité Universitätsmedizin Berlin - Campus Virchow Klinikum, Berlin
  - University of Heidelberg, Heidelberg
  - Ludwig-Maximilians-University, Munich
  - Klinikum rechts der Isar of the Technical University of Munich, Munich
- Hungary (2):
  - University of Pecs, Pécs
  - University of Szeged, Albert Szent Gyorgi Medical Center, Szeged

REFERENCES:
- [Background] Ward MD, Weber A, Merrill VD, Welch RD, Bazarian JJ, Christenson RH. Predictive Performance of Traumatic Brain Injury Biomarkers in High-Risk Elderly Patients. J Appl Lab Med. 2020 Jan 1;5(1):91-100. doi: 10.1093/jalm.2019.031393. PMID 32445344
- [Result] Bazarian JJ, Biberthaler P, Welch RD, Lewis LM, Barzo P, Bogner-Flatz V, Gunnar Brolinson P, Buki A, Chen JY, Christenson RH, Hack D, Huff JS, Johar S, Jordan JD, Leidel BA, Lindner T, Ludington E, Okonkwo DO, Ornato J, Peacock WF, Schmidt K, Tyndall JA, Vossough A, Jagoda AS. Serum GFAP and UCH-L1 for prediction of absence of intracranial injuries on head CT (ALERT-TBI): a multicentre observational study. Lancet Neurol. 2018 Sep;17(9):782-789. doi: 10.1016/S1474-4422(18)30231-X. Epub 2018 Jul 24. PMID 30054151
- [Derived] Bazarian JJ, Welch RD, Caudle K, Jeffrey CA, Chen JY, Chandran R, McCaw T, Datwyler SA, Zhang H, McQuiston B. Accuracy of a rapid glial fibrillary acidic protein/ubiquitin carboxyl-terminal hydrolase L1 test for the prediction of intracranial injuries on head computed tomography after mild traumatic brain injury. Acad Emerg Med. 2021 Nov;28(11):1308-1317. doi: 10.1111/acem.14366. Epub 2021 Sep 7. PMID 34358399